CLINICAL TRIAL: NCT05513547
Title: Beneficial Effects of Daytime Light Exposure and Physical Activity on the Human Circadian Clock and Sleep
Acronym: DayCiS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-01140; pk22Blume
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Circadian System
Keywords: daytime light exposure; human circadian clock; Dim-Light Melatonin Onset (DMLO); nocturnal light exposure; intrinsically photosensitive retinal ganglion cells (ipRGCs); retinal photoreceptors; photopic illuminance; melanopic illuminance; melanopic equivalent daylight illuminance (EDI)
MeSH Terms: interventions — P-2

STUDY DESIGN:
Intervention Model Description: Sequential Bayes Factor approach: spectral characteristics of daytime LE varied in a within-subject manner in three sequential 7-hour LE protocols (P1, P2, P3).
  Physical activity varied between subjects in two subgroups: one 'resting' group and one 'hiking' group. The latter will hike (P2/3) or walk on a treadmill (P1) for 4 hours during LE.
Masking Description: Blinding of participants and researchers is not possible in this design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- resting subgroup (Other): Will be allowed to engage in activities that do not require self-luminous displays (e.g., study/read, play boardgames, listen to podcasts) during the three scheduled 7-hour light exposure (LE) conditions. For 'resting' participants, the time they spend under the open sky, in the shade or half-shade, will be matched to what the 'hikers' experience.
  Interventions: Other: LE protocol 1: exposure to artificial light; Other: LE protocol 2: natural daylight; Other: LE protocol 3: natural daylight with reduced short-wavelength proportions
- hiking subgroup (Other): Will have 4 hours of scheduled moderate physical activity (average approx. 70-75% of maximum heart rate during each LE starting 3h after waking up to meet the circadian time when the most pronounced phase-advance is expected. The scheduled 4-hour activity will be a hike in the greater Basel area, which will cover about 12-14 km and a gain in elevation of less than 500 metres. Participants will be instructed to walk at their own speed. During protocol 1, which will take place in the lab, participants in the 'hiking' group will walk on a tiltable treadmill.
  Interventions: Other: LE protocol 1: exposure to artificial light; Other: LE protocol 2: natural daylight; Other: LE protocol 3: natural daylight with reduced short-wavelength proportions

INTERVENTIONS:
Other: LE protocol 1: exposure to artificial light — Participants stay in the lab with light mimicking usual office lighting. On days 8, 15, and 22, participants start the experimental protocol 5 hours before HBT: questionnaires, behavioural responsiveness (assessed by PVT), saliva samples for melatonin measurements (until HBT and two more following awakening the next day). Participants will go to bed at HBT and get up 8h later in the morning. Their sleep will be assessed with PSG recordings.
  Other Names: P1
Other: LE protocol 2: natural daylight — Participants spend the same time outdoors in natural daylight. On days 8, 15, and 22, participants start the experimental protocol 5 hours before HBT: questionnaires, behavioural responsiveness (assessed by PVT), saliva samples for melatonin measurements (until HBT and two more following awakening the next day). Participants will go to bed at HBT and get up 8h later in the morning. Their sleep will be assessed with PSG recordings.
  Other Names: P2
Other: LE protocol 3: natural daylight with reduced short-wavelength proportions — Participants spend the same time outdoors in natural daylight wearing tinted glasses that filter out short-wavelength light proportions. On days 8, 15, and 22, participants start the experimental protocol 5 hours before HBT: questionnaires, behavioural responsiveness (assessed by PVT), saliva samples for melatonin measurements (until HBT and two more following awakening the next day). Participants will go to bed at HBT and get up 8h later in the morning. Their sleep will be assessed with PSG recordings.
  Other Names: P3

SUMMARY:
This study is to examine the circadian phase-shifting effects of daylight and physical activity (primary endpoint: shift in dim-light melatonin onset (DLMO)) as well as their effects on sleep the ensuing night and analyzes how different spectral characteristics of daylight and physical activity affect the biological clock and sleep.

There are two types of interventions in a within-between study plan: - Within participants: light conditions will be varied during daytime in three 7-hour light exposure protocols (usual office lighting, natural daylight, natural daylight with "blue"-light filtering glasses). - Between participants: physical activity levels (rest vs. 4 hours of moderate activity, i.e., hiking) will be varied. Eligible volunteers are invited to partake in the three-week study schedule, including three experimental visits and in-between ambulatory sleep-wake and light exposure tracking. On study intake, participants are randomly assigned to either the 'hike' or 'rest' activity subgroup. The 'resting subgroup' will be allowed to study, read, etc. during the experimental conditions, whereas the 'hiking subgroup' will have 4 hours of scheduled moderate physical activity during each LE condition starting 3 hours after waking up.

Following the screening procedure and an adaptation night to screen for sleep disorders, eligible participants will be matched with a 'partner'. One will be assigned to the rest (A), the other to the hiking (B) subgroup. LE protocols within each subgroup are identical and participants from each pair will undergo all light conditions on the same day to minimize variability due to e.g., weather conditions.

DETAILED DESCRIPTION:
While phylogenetically, life on earth has developed under the cyclic changes of sunlight and darkness, human life in modern societies is usually characterized by a markedly different light environment: spending most of the waking day indoors in relatively low light levels, whereas exposing ourselves to relatively high levels of artificial light in the evening. This decrease in day-night contrast has detrimental effects on the human circadian system and sleep. The pathways that mediate these effects have functionally been mapped using evening or nocturnal light exposure (LE). It has been shown that light with increased short-wavelength proportions suppresses melatonin, delays the biological clock, and impairs sleep. These consequences are thought to be mainly mediated by the effects of short-wavelength light on intrinsically photosensitive retinal ganglion cells (ipRGCs), which express melanopsin that has its peak spectral sensitivity at around 480nm. Little is known about the contributions of the other retinal photoreceptors, particularly the cones, which encode colour and brightness under daylight viewing conditions. Thus, the precise contributions of melanopic and photopic illuminance remain to be established. Besides the negative effects of evening artificial LE, exposure to higher levels of daylight is associated with beneficial consequences for sleep and circadian rhythms. However, also in this respect, the precise photopic and melanopic contributions remain to be established. Beyond this, daylight exposure is often confounded with physical activity, which can act as a zeitgeber itself. Specifically, physical activity in the morning and the afternoon has been shown to acutely phase-advance the biological clock and positively affect sleep. The possible contributions of an interaction with LE remain to be established. This study aims at delineating the effects of (i) photopic and melanopic illuminance during daytime LE and (ii) physical activity on the biological clock and sleep. The spectral characteristics of daytime LE will be varied in a within-subject manner in three 7-hour LE protocols. Physical activity will be varied between subjects in two subgroups (i.e., 'hike' and 'rest'). This study investigates the relative importance of daytime and its precise spectral characteristics as well as physical activity for healthy circadian rhythms and sleep.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-35 years
* Body Mass Index: 18.5-24.9 (i.e., normal weight according to World Health Organization (WHO) criteria)
* Moderate cardiorespiratory fitness levels, moderate level of endurance training according to the category "moderate physical activity" (category 2) of the International Physical Activity Questionnaire (IPAQ) short form
* Informed consent as documented by signature of the participant

Exclusion Criteria:

* Self-reported pregnancy
* Investigator's family members, employees, or other dependent persons
* Chronic or debilitating medical (including psychiatric) conditions; normal state of health will be established on the basis of questionnaires and the examination by the physician in charge. Illnesses that would be a reason for exclusion are:

  * Sleep disorders: Narcolepsy, sleep apnea (apnea index > 10), periodic limb movements (PLM index > 15), insomnia (polygraphically recorded sleep efficiency < 70% or Pittsburgh Sleep Quality Index (PSQI) index > 5), hypersomnia
  * Chronobiological disorders: hypernychthemeral sleep-wake cycle, delayed or advanced sleep phase syndrome
  * Psychiatric disorders
  * Somatic diseases: cardiovascular, respiratory, gastrointestinal, haemopoietic, visual and immune system diseases, neurological disorders, infectious diseases, allergies (e.g., skin allergies, acute hay fever), thrombocytopenia or other dysfunctions of blood platelets
* Drug use: volunteers must not consume any drugs (including nicotine and alcohol) for the entire duration of the study with no history of drug or alcohol dependency. This will be ensured by the use of a urine multi-drug screen at every experimental visit.
* Medication that could affect outcome parameters
* Shift work < 3 months prior to study intake
* Transmeridian travel (> 2 time zones) < 1 month prior to study intake
* Extreme chronotype (Munich Chronotype Questionnaire [MCTQ] <2 or >7)
* Extremely long/short sleep duration (subjective sleep duration on workdays outside 6-10h according to the MCTQ)
* Abnormal colour vision, vision disorders (other than e.g., mild myopia corrected with contact lenses)
* Inability to understand and/or follow procedures
* Non-adherence to the circadian stabilization protocol during the five days prior to and between the experimental visits (deviation of >30min form scheduled times more than twice or on the day of the study visit)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Difference in salivary DLMO (in minutes, phase advance) between the first and the second night (Shift in dim-light melatonin onset (DLMO)) | On the evenings of each LE protocol (from 5 hours before habitual bedtime (HBT) (every 30 minutes)) and in the mornings during the first hour after wake-up (8h later) on day 8-10, day 15-17, day 22-24.
  Phase shift in the dim-light melatonin onset (DLMO) due to the light exposure from evening 1 to evening 2 of each experimental visit

SECONDARY OUTCOMES:
EEG slow-wave activity (SWA) (i.e., delta power density between 0.5 and 4.5 Hz) as an indicator of sleep propensity within each NREM part of a sleep cycle | On day 8-10, day 15-17, day 22-24.
  EEG SWA for each decile of the NREM part of the first non-rapid eye movement (NREM)-REM cycle will be computed. For the computation of delta power density, artefact-free data will be segmented into 2-second time bins and subjected to Fast Fourier Transformation (FFTs) yielding a frequency resolution of 0.5 Hz. Thereafter, FFT results will be averaged in the 0.5-4.5 Hz range at frontal electrodes F3, Fz, and F4 within each percentile of each NREM cycle. For each NREM cycle, the analyses will thus yield 10 measures per participant.
Change in Karolinska Sleepiness Scale (KSS) for subjective sleepiness | On the evenings of each LE protocol, from 5 hours before HBT on day 8-10, day 15-17, day 22-24.
  KSS is a single-item 9-point subjective Likert-type measurement scale for sleepiness
Change in Visual Comfort Scale (VCS) for mood, visual comfort and physical well-being. | On the evenings of each LE protocol, from 5 hours before HBT on day 8-10, day 15-17, day 22-24.
  Change in Visual Comfort Scale (VCS) to assess participants' mood, visual comfort and physical well-being under the different lighting conditions
Change in Psychomotor Vigilance Task (PVT) for objective alertness | On the evenings of each LE protocol, from 5 hours before HBT on day 8-10, day 15-17, day 22-24.
  Objective alertness will be measured using an acoustic version of the Psychomotor Vigilance Task (PVT). The test will run for a total of 10 min, stopping with the last response within this time frame. False starts will be coded for RTs <100 ms and lapses will be coded for RTs ≥ 2x median. After a response, the next tone will be played randomly after 2-10 s. The reaction time data will focus on mean 1/reaction time (mean 1/RT). Mean 1/RT will be calculated after the removal of false starts and lapses.
Change in Self-Assessment of Sleep and Awakening Quality Scale (SSA) for subjective sleep quality | Throughout the three weeks of the study protocol
  Sleep and wake episodes will be recorded using a sleep-wake diary (bedtime, lights-off, estimated sleep onset latency, number of waking up during night, number of getting up during night, wake-up time (lights-on), and getup time in the morning, type of day (work or free), activity during the day, daylight exposure, naps, time without the actimetry device, medicine, caffeine, and alcohol). Sleep quality rated on a Likert scale (1 = very poor to 8 = very good).
Change in Polysomnography (PSG)-derived sleep stages and arousals according to the AASM Manual for the Scoring of Sleep and Associated Events for objective sleep quality | During the nights of each experimental protocol (on day 8-10, day 15-17, day 22-24).
  Scoring of Polysomnography (PSG)-derived sleep stages
Change in actimetry (sleep-wake schedules) measured by actimetry devices | Throughout the three weeks of the study protocol
  Change in actimetry (sleep-wake schedules) by actimetry devices
Change in participants' light exposure, measured by lightweight light sensor | Throughout the three weeks of the study protocol
  Ambulatory light exposure will be assessed with a lightweight light sensor

CONTACTS AND LOCATIONS:
Overall Officials: Christine Blume, Dr. med., Principal Investigator — Centre for Chronobiology, Psychiatric Hospital of the University of Basel
Locations (1):
- Centre for Chronobiology, Psychiatric Hospital of the University of Basel, Basel, Switzerland